CLINICAL TRIAL: NCT03872648
Title: TransCare - Genital Surgery for Trans Women in Centralized vs. Decentralized Health Care Delivery Settings
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: TransCare2019
Record Dates: First submitted 2019-02-21; First posted 2019-03-13 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Gender Dysphoria; Gender Identity Disorder; Transsexualism; Gender Identity
MeSH Terms: conditions — Gender Dysphoria; Transsexualism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TW-VP (centralized delivery structure): Trans women seeking penile inversion vaginoplasty (TW-VP) assessing THC in a specialized clinic with a centralized structure
- TW-VP (decentralized delivery structure): Trans women seeking penile inversion vaginoplasty (TW-VP) assessing THC from different medical locations (decentralized structure)

SUMMARY:
Trans (i.e., transgender, transsexual) individuals experience a gender that does not match their sex assigned at birth (Gender Incongruence), which can lead to distress called gender dysphoria (formerly known as transsexualism). Trans health care (THC) is primarily focusing on transition-related medical interventions (e.g. genital surgery) to reduce gender dysphoria and improve the quality of life. To date, trans individuals access THC services in both decentralized (e.g., various transition-related interventions are spread over several locations) and centralized structures (e.g., gender affirmative medical treatments are provided by a single source). The TransCare study examines genital surgery for trans women (e.g. penile inversion vaginoplasty), focusing on the effect of different health care delivery settings (e.g., if patients received all treatments from a single source or spread over several locations) on psychosocial outcomes and the quality of healthcare.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years or older;
* Gender different from their assigned male sex at birth
* Current or new surgical care patient at Department of Urology at the University Medical Center Hamburg-Eppendorf
* Able to read, speak, and understand German
* Written informed consent after written and oral information

Exclusion Criteria:

* Under 16 years of age
* Missing informed consent
* Unable to speak German

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Eligible participants must identify with a gender different from their male sex assigned at birth
Study Population: Trans woman seeking for surgical care at the Department of Urology at the University Medical Center Hamburg-Eppendorf
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2019-01-21 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Gender Dysphoria (1) | Change from Baseline Gender Dysphoria to the point of time after penile inversion vaginoplasty (Baseline + 6 months) and to the 12 month post-procedure time point (Long-term-follow-up, Baseline +18 month)
  Gender Dysphoria is measured using the Transgender Congruence Scale (TCS; Kozee et al., 2012).
  The total scale score is calculated by averaging the responses of the items.
  Scaling: 1 (strongly disagree), 2 (somewhat disagree), 3 (neither agree nor disagree), 4 (somewhat agree); 5 (strongly agree)
  References:
  Kozee, H. B., Tylka, T. L., & Bauerband, L. A. (2012). Measuring transgender individuals' comfort with gender identity and appearance: Development and validation of the Transgender Congruence Scale. Psychology of Women Quarterly, 36(2), 179-196.
Gender Dysphoria (2) | Change from Baseline Gender Dysphoria to the point of time after penile inversion vaginoplasty (Baseline + 6 months) and to the 12 month post-procedure time point (Long-term-follow-up, Baseline +18 month)
  Gender Dysphoria is measured using the Gender Congruence and Life Satisfaction Scale (GCLS; Jones et al., 2018). A higher score indicates a more positive outcome.
  Scaling: 1 (Never), 2 (Rarely), 3 (Sometimes), 4 (Often), 5 (Always)
  References:
  Jones, B. A., Bouman, W. P., Haycraft, E., & Arcelus, J. (2018). The Gender Congruence and Life Satisfaction Scale (GCLS): Development and validation of a scale to measure outcomes from transgender health services. International Journal of Transgenderism, 1-18.
Quality of Life (physical health, psychological health, social relationships, and environment) | Change from Baseline QoL to the point of time after penile inversion vaginoplasty (Baseline + 6 months) and to the 12 month post-procedure time point (Long-term-follow-up, Baseline +18 month)
  QoL is measured using the WHOQOL-BREF (WHO, 1998).
  Reference:
  WHO (1998). Development of the World Health Organization WHOQOL-BREF quality of life assessment. Psychological medicine, 28(3), 551-558.
General symptoms related to mental health | Change from Baseline Mental Health Symptoms to the point of time after penile inversion vaginoplasty (Baseline + 6 months) and to the 12 month post-procedure time point (Long-term-follow-up, Baseline +18 month)
  General symptoms related to mental health are measured using the Basic Symptom Checklist (BSCL; Franke, 2015), which is the German version of the BSI-18.
  Reference:
  Franke, G. H. (2015). BSCL-53®-S. Brief Symptom-Checklist-Standard-Deutsches Manual.
Sexuality | Change from Baseline Sexuality to the point of time after penile inversion vaginoplasty (Baseline + 6 months) and to the 12 month post-procedure time point (Long-term-follow-up, Baseline +18 month)
  Sexuality (desire, arousal, lubrication, orgasm, satisfaction, and pain) is measured using the German Female Sexual Function Index (FSFI; Berner et al., 2004).
  Reference:
  Berner, M. M., Kriston, L., Zahradnik, H. P., Härter, M., & Rohde, A. (2004). Überprüfung der Gültigkeit und Zuverlässigkeit des deutschen Female Sexual Function Index (FSFI-d). Geburtshilfe und Frauenheilkunde, 64(03), 293-303.

SECONDARY OUTCOMES:
Patient-Centeredness | After the first stage of penile inversion vaginoplasty (Baseline + 2 weeks), after the second stage of penile inversion vaginoplasty (Baseline + 6 months)
  Five dimensions of patient-centredness (according to Scholl et al., 2014)
  1. Patient as a unique person
  2. Patient involvement in care
  3. Patient information
  4. Clinician-patient communication
  5. Patient empowerment
  Reference:
  Scholl, I., Zill, J. M., Härter, M., & Dirmaier, J. (2014). An integrative model of patient-centeredness-a systematic review and concept analysis. PloS one, 9(9), e107828.

CONTACTS AND LOCATIONS:
Overall Officials: Timo Nieder, Dr. phil., Principal Investigator — University Medical Center Hamburg-Eppendorf, Institute for Sex Research, Sexual Medicine and Forensic Psychiatry; Peer Briken, Prof., Study Director — University Medical Center Hamburg-Eppendorf, Institute for Sex Research, Sexual Medicine and Forensic Psychiatry
Locations (1):
- University Medical Center Hamburg-Eppendorf, Institute for Sex Research, Sexual Medicine and Forensic Psychiatry, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided